CLINICAL TRIAL: NCT05824637
Title: Validation and Reproducibility of Type I Hypersensitivity Reaction in the Diagnostic Process of the Skin Prick Test in Allergic and Non-allergic Individuals
Brief Title: Validation and Reproducibility of S.P.A.T. With Allergens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hippocreates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1794559
Record Dates: First submitted 2023-01-30; First posted 2023-04-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-07

CONDITIONS: Allergy to House Dust; Allergy Pollen
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin Prick Test (Other): Study participants will receive a skin prick test by the skin prick automated test device on the right arm and manually by a health care provider on the left arm.
  Interventions: Device: Skin Prick Automated Test; Diagnostic Test: Skin Prick Manual Test

INTERVENTIONS:
Device: Skin Prick Automated Test — skin prick test to detection sensitisation to aeroallergens
Diagnostic Test: Skin Prick Manual Test — skin prick test to detection sensitisation to aeroallergens

SUMMARY:
To improve accuracy and take out human error opportunities, Hippo Dx developed S.P.A.T., an automated skin prick test. This study will provide a comparison between manual and automated skin prick test in allergic and non-allergic individuals with a panel of common inhalant allergens.

The primary endpoint is to compare the accuracy of S.P.A.T. to detect sensitization to common aeroallergens compared to a manual skin prick test (SPT).

It is a prospective monocentric study that will include 120 study participants.

ELIGIBILITY:
Inclusion Criteria:

Adults (18-65y) with presence or absence of self-reported symptoms of inhalant allergy will be included.

Exclusion Criteria:

* Skin pathology like chronic or exuberant urticaria, dermographism, chronic dermatitis that needs daily treatment
* Use of antihistaminic medication < 7 days before the start of the study
* Use of tricyclic antidepressants (antihistamine activity) < 7 days before the start of the study
* Use of topical corticoids on the forearm < 7 days before the start of the study
* Use of Omalizumab < 6 months before the start of the study
* Pregnancy: there is a remote possibility of inducing a systemic allergic reaction that could induce uterine contractions or necessitate the use of epinephrine (thought to cause constriction of the umbilical artery)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Within-test agreement (% of patients with consistent results) of wheal positivity per allergen between manual and automated test. | 15 minutes after the diagnostic test
  Each of the allergens are pricked three times via manual and automated skin prick test. Three positive or negative test results are considered consistent whereas either one or two positive or negative test results are considered non-consistent resulting in an inconclusive test result.

SECONDARY OUTCOMES:
Allergy symptoms assessed by visual analogue scale between patients with a positive versus negative test result. | day of the diagnostic test
  Visual analogue scale (0: best - 10: worse)
Time (seconds) required to run an automated versus a manual skin prick test. | during the diagnostic test
Amount of allergen solution that is required to run an automated versus a manual skin prick test. | during the diagnostic test
Level of discomfort experienced by the patient as assessed by visual analogue scale after an automated versus a manual skin prick test. | 15 minutes after the diagnostic test
  Visual analogue scale (0: best - 10: worse)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Sebrechts, MD, Principal Investigator — AZ Herentals
Locations (1):
- AZ Herentals, Herentals, Belgium

IPD SHARING:
Plan to Share IPD: No